CLINICAL TRIAL: NCT06765252
Title: Effect of Genetic Polymorphism on Capecitabine-Induced Toxicity in Egyptian Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Principal Investigator, Raghad Essam Nassar, Teaching Assistant, Clinical Pharmacy Department, Faculty of Pharmacy, Menoufia University, Menoufia University
Other Study IDs: 4/2024ONCO16; 281 (Other: Faculty of Pharmacy Ain Shams University)
Record Dates: First submitted 2024-11-12; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer; Breast Cancer
Keywords: Polymorphism; CES1; Capecitabine; Toxicity; Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Capecitabine-based chemotherapy — Participants receiving capecitabine in an oral dose of 1,000-1,250 mg/m2 twice daily for the first 14 days of each 21-day cycle.

SUMMARY:
The goal of this observational study is to study the effect of a single nucleotide polymorphism in the CES1 gene (rs2244613) on capecitabine-induced toxicity in Egyptian cancer patients. This study will help in understanding the interindividual variability in the CES1 gene and the effect of a single nucleotide polymorphism in this gene (rs2244613) on capecitabine-induced toxicity in participants already taking capecitabine-based chemotherapy as part of their regular medical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast or colorectal cancer receiving capecitabine-based chemotherapy
* Age > 18 years
* ECOG PS 0-2.

Exclusion Criteria:

* Patients treated with irinotecan
* Lack of physical integrity of the upper gastrointestinal tract
* Patients with malabsorption syndrome
* Patients having inability to take oral medication
* Patients with poor performance status
* Patients with chronic diarrhea as ulcerative colitis or Crohn's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Egyptian cancer patients presenting to the department of Clinical Oncology, Faculty of Medicine, Menoufia University.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of gastrointestinal toxicity | Six months
  Occurrence and severity of capecitabine-induced gastrointestinal toxicity will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE V5.0) in relation to the variation in patients' genotype of rs2244613 in the CES1 gene.
Occurrence of hand-foot syndrome | Six months
  Occurrence and severity of capecitabine-induced Hand-foot syndrome will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE V5.0) in relation to the variation in patients' genotype of rs2244613 in the CES1 gene.

SECONDARY OUTCOMES:
Occurrence of hematological toxicity | Six months
  Occurrence and severity of capecitabine-induced hematological toxicity will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE V5.0) in relation to the variation in patients' genotype of rs2244613 in the CES1 gene.
Occurrence of hepatic toxicity | Six months
  Occurrence and severity of capecitabine-induced hyperbilirubinemia will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE V5.0) in relation to the variation in patients' genotype of rs2244613 in the CES1 gene.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Faculty of Medicine, Menoufia University, Shibīn al Kawm, Menoufia, Egypt